CLINICAL TRIAL: NCT02661594
Title: A Randomised, Double-blind, Four-period Crossover Study to Investigate the Effect of Intravenous APD421 on Cardiac Conduction as Compared to Placebo and Moxifloxacin in Healthy Adult Subjects
Brief Title: Thorough QT Study of Intravenous Amisulpride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: DP10013
Record Dates: First submitted 2016-01-14; First posted 2016-01-22 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: TQT; amisulpride; volunteer; ECG
MeSH Terms: interventions — Amisulpride; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ABCD (Experimental): A: APD421 5 mg followed by B: APD421 40 mg; C: Moxifloxacin 400 mg; D: Placebo.
  Interventions: Drug: APD421 5 mg; Drug: APD421 40 mg; Drug: Moxifloxacin; Drug: Placebo
- BDAC (Experimental): B: APD421 40 mg; D: Placebo. A: APD421 5 mg C: Moxifloxacin 400 mg;
  Interventions: Drug: APD421 5 mg; Drug: APD421 40 mg; Drug: Moxifloxacin; Drug: Placebo
- CADB (Experimental): C: Moxifloxacin 400 mg A: APD421 5 mg D: Placebo B: APD421 40 mg
  Interventions: Drug: APD421 5 mg; Drug: APD421 40 mg; Drug: Moxifloxacin; Drug: Placebo
- DCBA (Active Comparator): D: Placebo C: Moxifloxacin 400 mg B: APD421 40 mg A: APD421 5 mg
  Interventions: Drug: APD421 5 mg; Drug: APD421 40 mg; Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: APD421 5 mg — Therapeutic dose of amisulpride
  Other Names: Amisulpride 5mg
Drug: APD421 40 mg — Supra-therapeutic dose of amisulpride
  Other Names: Amisulpride 40mg
Drug: Moxifloxacin — Positive control for assay sensitivity
Drug: Placebo — Placebo comparator to establish baseline for calculating change in QTcF

SUMMARY:
Randomised, single-dose, crossover, placebo-controlled study to see if intravenous amisulpride has any effect on the heart rhythm, in particular the QT interval, in healthy adult volunteers.

DETAILED DESCRIPTION:
Phase 1, randomised, single-dose, period-balanced, crossover, placebo- controlled study to assess the effects of iv doses of amisulpride on the QT interval, corrected for heart rate by Fridericia's formula (QTcF), in healthy male and female subjects of Caucasian and Japanese ethnicity aged 20-45 years.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged between 20 and 45 years (inclusive) at screening.
2. Signed informed consent in the local language prior to any study-mandated procedure.
3. Japanese subjects defined as a person carrying a Japanese passport, who is a descendant of four Japanese grandparents and has not been outside Japan for more than five years prior to screening.
4. The Caucasian subjects should be distinguished especially by very light to brown skin pigmentation and straight to wavy or curly hair, and should be indigenous to Europe, northern Africa, western Asia, and India. Therefore, the study may as well include Caucasian subjects from North America, Australia and South Africa
5. No clinically significant findings on the physical examination at screening and at admission on Day -2.
6. Body mass index (BMI) between 18 and 25 kg/m2 (inclusive) at screening and at admission on Day -2, body weight at least 48 kg.
7. Systolic blood pressure (SBP) 90-145 mmHg, diastolic blood pressure (DBP) 40-90 mmHg, and heart rate (HR) 40-90 bpm (all inclusive), measured on the left arm, after 10 minutes in the supine position at screening and at admission on Day -2.
8. Triplicate 12-lead ECG without clinically relevant abnormalities measured after ten minutes in the supine position at screening and on admission on Day -2.
9. 24-hour 12-lead Holter ECG or an equivalent assessment and/or submaximal exercise test without clinically relevant abnormalities measured at screening.
10. Haematology, biochemistry and urinalysis test results not deviating from the normal range to a clinically relevant extent at screening and at admission.
11. Subjects must agree to use acceptable methods of contraception:

    Male subjects

    Male subjects must use medically acceptable methods of contraception if their female partner(s) is (are) pregnant or lactating from the time of the first administration of treatment or study medication until three months following administration of the last treatment or dose of study medication. Acceptable methods include:
    * Condom used with spermicidal foam/gel/film/cream/suppository
    * If the subject has undergone surgical sterilisation (vasectomy with documentation of azoospermia) a condom with spermicidal foam/gel/film/cream/suppository must be used.

    Use acceptable methods of contraception if the male subject's partner could become pregnant from the time of the first administration of treatment or study medication until three months following administration of the last treatment or dose of study medication. The acceptable methods of contraception are as follows:
    * Condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
    * Surgical sterilisation (vasectomy with documentation of azoospermia) and a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps] used with spermicidal foam/gel/film/cream/suppository).
    * The female partner uses oral contraceptives (combination oestrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps] used with spermicidal foam/gel/film/cream/suppository).
    * The female partner uses medically prescribed topically-applied transdermal contraceptive patch and a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps] used with spermicidal foam/gel/film/cream/suppository).
    * The female partner has undergone documented tubal ligation (female sterilisation). In addition, a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps] used with spermicidal foam/gel/film/cream/suppository) must be used.
    * The female partner has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS) and the use of a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps] used with spermicidal foam/gel/film/cream/suppository).
    * True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

    Female subjects

    Female subjects of childbearing potential must use medically acceptable methods of contraception from the time of the first administration of treatment or study medication until three months following administration of the last treatment or dose of study medication. Acceptable methods include:
    * A documented placement of an IUD or IUS and the use of a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps) used with spermicidal foam/gel/film/cream/suppository]).
    * Documented tubal ligation (female sterilisation). In addition, a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps] used with spermicidal foam/gel/film/cream/suppository) should also be used.
    * Double barrier method: Condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
    * True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) are not acceptable methods of contraception.
12. Ability to communicate well with the Investigator in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Women who are pregnant and/or breastfeeding.
2. Received amisulpride for any indication within the last 2 weeks.
3. Allergy to amisulpride or any of the excipients of APD421.
4. History of vestibular disorder or history of dizziness.
5. Received anti-emetic therapy including corticosteroids within the last 2 weeks.
6. History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study drug (appendectomy and herniotomy allowed, cholecystectomy not allowed).
7. History of epilepsy.
8. History of clinically significant syncope.
9. Family history of sudden death.
10. Family history of premature cardiovascular death.
11. Clinically significant history or family history of congenital long QT syndrome (e.g. Romano-Ward syndrome, Jervell and Lange-Nielson syndrome) or Brugada's syndrome.
12. History of clinically significant arrhythmias and ischemic heart disease (especially ventricular arrhythmias, atrial fibrillation (AF), recent conversion from AF or coronary spasm).
13. Conditions predisposing the volunteer to electrolyte imbalances (e.g. altered nutritional states, chronic vomiting, anorexia nervosa, bulimia nervosa).
14. ECG abnormalities in the standard 12-lead ECG (at screening and Day -2) and 24-hour 12-lead Holter ECG or an equivalent assessment and/or submaximal exercise test (at screening) which in the opinion of the Investigator will interfere with the ECG analysis.
15. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes. This includes subjects with any of the following (at screening and Day -2 of Period 1):

    * Sinus node dysfunction.
    * Clinically significant PR (PQ) interval prolongation.
    * Intermittent second or third degree atrioventricular (AV) block.
    * Incomplete or complete bundle branch block.
    * Abnormal T-wave morphology.
    * Prolonged QT interval corrected with Bazett's formula (QTcB) >450 ms or shortened QTcB < 350 ms or family history of long QT syndrome.

    Subject with borderline deviations from these criteria may be included if the deviations do not pose a safety risk, and if agreed between the appointed Cardiologist and the PI.
16. Signs and/or symptoms of a clinically relevant acute illness in the four-week period prior to screening.
17. Veins unsuitable for intravenous puncture or cannulation on either arm (e.g. veins that are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture).
18. Known hypersensitivity to any medicines administered in the trial.
19. Treatment with any prescribed medication during the two weeks prior to first baseline day.
20. Treatment with any over-the-counter (OTC) medications during the two weeks prior to first baseline day.
21. Treatment with vitamins and/or minerals within 48 hours prior to the first baseline day.
22. Treatment with another investigational drug within four weeks prior to dosing or having participated in more than three investigational drug studies within one year prior to dosing.
23. Confirmed positive results from urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates and methadone) or from the alcohol breath test at screening and on Day -2.
24. History or clinical evidence of alcoholism or drug abuse. Alcohol abuse is defined as regular weekly intake of more than 14 units (Using alcohol tracker http://www.nhs.uk/Tools/Pages/NHSAlcoholtracker.aspx); drug abuse is defined as compulsive, repetitive and/or chronic use of drugs or other substances with or without problems related to their use and/or where stopping or a reduction in dose will lead to withdrawal symptoms.
25. Excessive caffeine consumption, defined as ≥800 mg per day at screening (800 mg = 7 cups of coffee or 16 cups of tea).
26. Smoking within three months prior to screening or during the screening period.
27. Loss of 250 mL or more blood within three months prior to screening.
28. Positive results from the hepatitis serology, except for vaccinated subjects, at screening.
29. Positive results from the HIV serology at screening.
30. Any circumstances or conditions, which, in the opinion of the Investigator, may affect full participation in the study or compliance with the protocol.
31. Legal incapacity or limited legal capacity at screening.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Fox, MB BChir, Study Director — Acacia Pharma Ltd

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty (40) healthy, non-elderly, Caucasian and Japanese, male or female subjects were planned to enter the study. At least 10 subjects were to be Japanese and at least 40% of subjects for both races were to be male.
Pre-assignment Details: Forty (40) healthy subjects entered the study. One subject voluntarily withdrew after Period 1 (moxifloxacin 400 mg) and another subject was withdrawn due to severe non-compliance with the protocol after receiving APD421 5 mg and 40 mg.
Groups:
- BDAC: B: APD421 40 mg; D: Placebo. A: APD421 5 mg C: Moxifloxacin 400 mg.
Period: Overall Study
Arm/Group | ABCD | BDAC | CADB | DCBA
Started | 10 | 11 | 10 | 9
Completed | 9 | 11 | 9 | 9
Not Completed | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABCD | BDAC | CADB | DCBA | Total
Number analyzed (Participants) | 10 | 11 | 10 | 9 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.50 (4.22) | 26.82 (4.24) | 30.20 (8.07) | 27.44 (4.93) | 27.99 (5.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 4 | 17
  Male | 6 | 6 | 6 | 5 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 4 | 4 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 5 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximal Mean ΔΔQTcF
Description: Maximal mean placebo-corrected change from baseline of QTcF (QT interval corrected for heart rate using the Fridericia formula) for single 5 mg and 40 mg iv doses of APD421. At each time point (2 mins, 8 mins, etc) the QTcF is compared to the pre-dosing "baseline" value, in order to calculate the change in QTcF (ΔQTcF). The value of ΔQTcF at each time point is then compared against the same time point for a placebo infusion, and the difference is calculated (ΔΔQTcF).
Time Frame: 24 hours
Measure: Mean (90% Confidence Interval); unit: milliseconds
Groups:
- 5 mg IV APD421: Single dose of 5 mg IV APD421 infused over 2 minutes
- 40 mg IV APD421: Single dose of 40 mg IV APD421 infused over 2 minutes
- Placebo: IV placebo infused over 8 minutes
- Oral Moxifloxacin: Single 400 mg oral dose of moxifloxacin
Arm/Group | 5 mg IV APD421 | 40 mg IV APD421 | Placebo | Oral Moxifloxacin
Number analyzed (Participants) | 39 | 39 | 38 | 39
milliseconds | 5.0 [2.8 to 7.1] | 23.4 [21.3 to 25.5] | 0.8 [-1.4 to 2.9] | 12.3 [10.1 to 25.5]

ADVERSE EVENTS:
Time Frame: All AE's are to be reported within a timeframe of 24hours.
Description: All AE encountered during the study will be reported in detail in the source documents and noted in the AE section of the CRF from the date of subject consent, throughout the clinical conduct and up to the follow-up visit. for a period of 24hours
Groups:
- Placebo: Intravenous placebo: two infusions in parallel, one over 2 minutes, one over 8 minutes
  Placebo: Placebo comparator to establish baseline for calculating change in QTcF
- Amisulpride 5 mg: Intravenous amisulpride 5 mg: infusion over 2 minutes; Intravenous placebo infused in parallel over 8 minutes
  Amisulpride 5 mg: Therapeutic dose of amisulpride
- Amisulpride 40 mg: Intravenous amisulpride 40 mg: infusion over 8 minutes;
  Intravenous placebo infused in parallel over 2 minutes
  Amisulpride 40 mg: Supra-therapeutic dose of amisulpride
- Moxifloxacin: Oral moxifloxacin 400 mg tablet administered once (not blinded)
  Moxifloxacin: Positive control for assay sensitivity
Arm/Group | Placebo | Amisulpride 5 mg | Amisulpride 40 mg | Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39 | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 9/38 | 5/39 | 35/39 | 5/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=38) | Amisulpride 5 mg (N=39) | Amisulpride 40 mg (N=39) | Moxifloxacin (N=39)
Infusion-related reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 20 (20) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Application site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Infusion Site Pain (General disorders) | 1 (1) | 0 (0) | 7 (8) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
There were no limitations and caveats with this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days